CLINICAL TRIAL: NCT04412577
Title: A Phase I, Open-label, Dose Escalation and Expansion Study to Evaluate the Tolerance, Efficacy and Pharmacokinetics of TQB3473 Tablets
Brief Title: A Study of TQB3473 Tablets in Subjects With Relapsed or Refractory Hematological Malignancies
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB3473-I-01
Record Dates: First submitted 2020-05-28; First posted 2020-06-02 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Relapsed/Refractory Hematological Malignancies
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB3473 tablets (Experimental): TQB3473 tablets administered once daily in 28-day cycle .
  Interventions: Drug: TQB3473

INTERVENTIONS:
Drug: TQB3473 — TQB3473 tablets administered orally once. Then TQB3473 tablets administered orally, once daily in 28-day cycle after 3 days of first administration.

SUMMARY:
This is a study to evaluate the maximum tolerated dose (MTD), occurrence of all adverse events (AE) and serious adverse events (SAE) , pharmacokinetic parameters and antitumor effect of TQB3473 tablets in Chinese adult patients with Relapsed or refractory hematological malignancies.

ELIGIBILITY:
Inclusion Criteria:

-1.Understood and signed an informed consent form. 2. Relapsed or refractory malignant hematological tumors. 3. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 1; Life expectancy ≥12 weeks.

4. Has at least one measurable lesion. 5. Adequate organ system function. 6. Patients need to adopt effective methods of contraception.

Exclusion Criteria:

* 1. Severe hypersensitivity to the drug or ingredients. 2. Has received chemotherapy, radiotherapy, immunotherapy or any other anti-tumor therapy within 14 days before the first dose.

  3. Has received spleen tyrosine kinase (SYK) inhibitors. 4. Has to use ≥ 10 mg/day glucocorticoid prednisone. 5. Has received BTK inhibitors and PI3K inhibitors before the first dose. 6. Has received allogeneic hematopoietic stem cell transplantation. 7. Has received autologous hematopoietic stem cell transplantation within 12 weeks before the first dose.

  8. Has any acute or chronic gastrointestinal diseases. 9. Has primary central nervous system lymphoma, or brain metastases with clinical symptoms, spinal cord compression, cancerous meningitis.

  10. Intermediate-risk or high-risk myelodysplastic syndrome. 11. Pregnancy and lactation women. 12. Has any serious and/or uncontrollable disease. 13. Has active autoimmune disease and received immunosuppressive therapy. 14. Has a history of neurological or mental disorders. 15. Has uncontrollable systemic bacterial, fungal or viral active infections 16. The toxicity of previous antitumor treatment is not recovered to ≤ grade 1. 17. Has other malignancies. 18. Has received surgery within 4 weeks before the first administration. 19. Has participated in any other clinical trials. 20. According to the judgement of the investigators, there are other factors that may lead to the termination of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2020-10-12 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | up to 31 days
  MTD was defined as the dose in which more than 2 of up to 6 patients developed a DLT.

SECONDARY OUTCOMES:
Tmax | 30minutes, 1hour, 2hour, 4hour, 6hour, 8hour,12hour, 24hour, 48hour post-dose on day 1 and day 31; 30minutes pre-dose on day 1, day 4, day 11,day 18 ,day 25 and day 31.
Cmax Cmax | 30minutes, 1hour, 2hour, 4hour, 6hour, 8hour,12hour, 24hour, 48hour post-dose on day 1 and day 31; 30minutes pre-dose on day 1, day 4, day 11,day 18 ,day 25 and day 31.
AUC0-t | 30minutes, 1hour, 2hour, 4hour, 6hour, 8hour,12hour, 24hour, 48hour post-dose on day 1 and day 31; 30minutes pre-dose on day 1, day 4, day 11,day 18 ,day 25 and day 31.
Overall response rate (ORR) | up to 96 weeks
  Percentage of subjects achieving complete response (CR) and partial response (PR).
Progression-free survival (PFS) | up to 96 weeks
  PFS defined as the time from first dose to the first documented progressive disease (PD) or death from any cause.
Duration of Response (DOR) | up to 96 weeks
  DOR defined as time from earliest date of disease response to earliest date of disease progression based on radiographic assessment.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality